CLINICAL TRIAL: NCT04036838
Title: ARJ C13 Urea Breath Test System
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ARJ Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ARJ 2014-01
Record Dates: First submitted 2019-07-25; First posted 2019-07-30 (Actual); Results first posted 2019-10-02 (Actual); Last update posted 2019-10-23 (Actual); Status verified 2019-10

CONDITIONS: H. Pylori Infection
MeSH Terms: interventions — Shadowing Technique, Histology

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Indication for H.pylori testing (Experimental): Walk in basis: Symptomatic patients of H.pylori infection will be enrolled for this study if all acceptance criteria are met. Patients will undergo C13 Urea Breath Test in addition to at least 2 other diagnostic tools from one obtained biopsy as comparison.
  Interventions: Combination Product: PyloPlus UBT System; Diagnostic Test: Histology; Diagnostic Test: Rapid Urease Test; Diagnostic Test: H.pylori Culture

INTERVENTIONS:
Combination Product: PyloPlus UBT System — Breath will be analyzed for change in carbon 13 content in breath after ingestion of enriched carbon 13 urea.
Diagnostic Test: Histology — Biopsy specimen fixed with 10% buffered formalin were cut into 4mm sections, stained with Giemsa stain, and examined by experienced pathologist
Diagnostic Test: Rapid Urease Test — Biopsy specimen obtained and placed onto Rapid Urease Test
Diagnostic Test: H.pylori Culture — Biopsy specimen obtained and sent to lab for culture analysis

SUMMARY:
An open-label, comparative group study to evaluate the equivalency of the PyloPlus 13C Urea Breath Test to predicate devices on the market.

DETAILED DESCRIPTION:
An open-label, comparative group study to evaluate the equivalency of the PyloPlus 13C Urea Breath Test to predicate devices on the market. Predicate devices include: Histology, Culture, RUT, and other 13C Breath Tests.

ELIGIBILITY:
Inclusion Criteria:

* Male or female at least 18 years of age at the time of visit
* Patients who are experiencing the effects of gastritis
* Written informed consent (and assent when applicable) obtained from subject and ability for subject to comply with the requirements of the study

Exclusion Criteria:

* Pregnant or lactating women.
* Study subjects currently taking antibiotics
* Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data
* Fasting required one hour prior to testing
* Study subjects shall not consume the following items prior to the test: Mouthwash, Chewing Gum, Carbonated Beverages, Cigarette Smoke, Acetone (to stimulate the effect of ketone production that may result from some diets), Alcohol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 415 (Actual)
Dates: Start 2015-07-06 (Actual); Primary Completion 2017-06-14 (Actual); Study Completion 2017-06-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - American Gastroenterology and Hepatology, Clearwater, Florida
  - South Lake Gastrenology, Clermont, Florida
  - Florida Center for Gastroenterology, Largo, Florida
  - Habana Medical Center, Tampa, Florida
  - Whitaker, Weintraub & Grizzard, Tampa, Florida
  - Bay Area Gastroenterology Associates, Trinity, Florida

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Indication for H.Pylori Testing
Started | 415
Completed | 324
Not Completed | 91

BASELINE CHARACTERISTICS:
Arm/Group | Indication for H.Pylori Testing
Number analyzed (Participants) | 324
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 203
  >=65 years | 121
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 220
  Male | 104
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 3
  Black or African American | 13
  Hispanic | 59
  Other/Unknown/Not Reported | 116
  White | 133
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 324

OUTCOME MEASURES:

1. Primary Outcome: Overall Percent Agreement
Description: The primary study endpoint is the performance measure in initial diagnosis (histology, RUT, culture) compared to the PyloPlus 13C UBT System
  Primary outcome of this study is to provide overall percent agreement in initial diagnosis with the PyloPlus 13C UBT System in comparison to other known diagnostic tools (histology, RUT, culture).
Time Frame: 2 Visits
Measure: Number (95% Confidence Interval); unit: percentage of pos. agreement
Arm/Group | Indication for H.Pylori Testing
Number analyzed (Participants) | 324
percentage of pos. agreement
  Sensitivity | 98.40 [91.7 to 99.7]
  Specificity | 99.20 [97.2 to 99.8]

ADVERSE EVENTS:
Time Frame: 2 Days
Arm/Group | Indication for H.Pylori Testing
All-Cause Mortality (participants affected / at risk) | 0/324
Serious Adverse Events (participants affected / at risk) | 0/324
Other Adverse Events (participants affected / at risk) | 0/324

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-06-26): https://cdn.clinicaltrials.gov/large-docs/38/NCT04036838/Prot_SAP_000.pdf